CLINICAL TRIAL: NCT05723432
Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Initial Efficacy of KD6001 in Combination With Anti-PD-1 Antibody in Patients With Advanced Melanoma
Brief Title: KD6001 in Combination With Anti-PD-1 Antibody in Patients With Advanced Melanoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Kanda Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KD6001CT02
Record Dates: First submitted 2023-02-03; First posted 2023-02-10 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — toripalimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KD6001+Toripalimab (Experimental): KD6001 combined with toripalimab in patients with advanced melanoma
  Interventions: Drug: KD6001; Drug: Toripalimab

INTERVENTIONS:
Drug: KD6001 — KD6001 will be administered intravenously.
Drug: Toripalimab — Toripalimab will be administered intravenously.
  Other Names: JS001

SUMMARY:
This is a phase 1b/2, open label study to evaluate the safety, tolerability, pharmacokinetics and initial efficacy of KD6001 in combination with toripalimab in patients with advanced melanoma.

ELIGIBILITY:
Main Inclusion Criteria:

1. Being voluntary to sign the informed consent form.
2. Male or female, aged ≥ 18 years.
3. Patients whose estimated survival time is more than 3 months.
4. Eastern Cooperative Oncology Group (ECOG) performance status score 0 or 1.
5. Histologically or cytologically confirmed advanced or metastatic melanoma, and the overall proportion of subjects with mucosal malignant melanoma will not exceed 22%.
6. At least one measurable lesion is used as the target lesion according to the Response Evaluation Criteria in Solid Tumors Version 1.1(RECIST V1.1).
7. The results of laboratory examination during the screening period suggest that the subjects have good organ function.
8. Male subjects with reproductive ability or female subjects with the possibility of pregnancy use effective contraceptive methods.
9. Good compliance and follow-up.

Main Exclusion Criteria:

1. Systematic treatment with antitumor drugs within 4 weeks prior to the start of this study.
2. Received immunotherapy (including PD-1/PD-L1 therapy and cell therapy) within 4 weeks prior to the start of this study.
3. Prior treatment with anti-CTLA-4 antibody.
4. Subjects with an active, known or suspected autoimmune disease.
5. Subjects with hepatitis (nonalcoholic steatohepatitis, alcoholic or drug-related, autoimmune hepatitis) and liver cirrhosis; active hepatitis B or hepatitis C.
6. Subjects with an active infection requiring systemic treatment.
7. Known history of testing positive for human immunodeficiency virus (HIV).
8. Subjects known to have active tuberculosis (TB).
9. Known to be allergic to KD6001 or Toripalimab and its components.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-03-22 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Dose Limiting Toxicities (DLTs) | Up to Day 21
  DLTs will be assessed during the dose-escalation phase and are defined as the following treatment-related adverse events occurring within a total of 21 days after the first trial administration.
The incidence and safety profile of participants with adverse events (AEs), serious adverse events(SAE), and immune-related adverse event(irAE) | Baseline to study completion up to 2 years
  Evaluate the adverse events (AE) according to National Cancer Institute Common Terminology Criteria for Adverse Events v5.0 (NCI CTCAE 5.0).
Maximum tolerated dose (MTD) | Up to Day 21
  The maximum tolerated dose (MTD) of KD6001 combined with toripalimab
Recommended Phase II dose (RP2D) | Up to Day 21
  Recommended Phase 2 dose (RP2D) of KD6001 combined with toripalimab

SECONDARY OUTCOMES:
The antitumor activity of KD6001 in combination with Toripalimab measured by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and modified RECIST 1.1 | Baseline to study completion up to 2 years
  Number of participants with response according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria and modified RECIST 1.1
The PK profile of KD6001 in combination with Toripalimab | Baseline to study completion up to 2 years
  Drug concentration of individual subject at different time points after administration; Pharmacokinetic parameters
The immunogenicity of KD6001 in combination with Toripalimab | Baseline to study completion up to 2 years
  Including the incidence of ADA positive. For ADA positive patients, the incidence of neutralizing antibody (NAB) will be analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, China